CLINICAL TRIAL: NCT00944567
Title: A Clinico-Pathologic Study of Primary Mediastinal B-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG26; EudraCT number 2006-005794-22
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Primary Mediastinal B-Cell Lymphoma
Keywords: Primary Mediastinal B-Cell Lymphoma; Positron emission tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
A non-profit study designed with the aim of analysing the phenotype and molecular characteristics (central review) and evaluating prospectively the role of PET-scans in the management of primary mediastinal lymphoma treated with conventional approaches.

ELIGIBILITY:
Inclusion Criteria:

* Primary mediastinal diffuse large B-cell lymphoma, CD20 positive. Patients must have histological confirmation of the diagnosis, and in addition have a dominant mass within the anterior mediastinum.
* No prior treatment of lymphoma. Patients may have received corticosteroids for up to 1 week for the relief of local compressive symptoms.
* Any stage of disease.
* Age at least 18 years.
* Fit to receive chemotherapy with curative intent.
* Able and willing to give informed consent, and to undergo staging including PET scanning
* Willingness to comply with an appropriate contraceptive method in women of childbearing potential or men.

Exclusion Criteria:

* Evidence of clinically significant cardiac disease, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months before study entry. Cardiac compromise due to local extension of lymphoma will not be an exclusion criterion in the absence of other cardiac disease.
* Impairment of bone marrow function (WBC <3.0x109/L, ANC <1.5x109/L, PLT <100x109/L), unless due to involvement by lymphoma.
* Major impairment of renal function (serum creatinine >2x upper normal) or liver function (ASAT/ALAT >2,5 upper normal, total bilirubin >2,5x upper normal), unless due to lymphoma involvement.
* Known HIV infection. Patients will not be tested routinely.
* Pregnant or lactating women.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient must have histological confirmation of the diagnodis of primary mediastinal diffuse large B cell lymphoma and have a dominant mass within the anterior mediastinum
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
response rate on PET scanning following initial chemo-immunotherapy

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (16):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - IRCCS Ospedale Oncologico, Bari
  - Policlinico S. Orsola Malpighi, Bologna
  - Ospedale Oncologico, Cagliari
  - Policlinico Careggi, Florence
  - A.O.Papardo, Messina
  - Ospedale Niguarda Ca' Granda, Milan
  - Ospedale San Raffaele, Milan
  - Università di Modena, Policlinico, Modena
  - Policlinico S. Matteo, Pavia
  - A.O. Bianchi-Melacrino-Morelli, Reggio Calabria
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Università di Roma "La Sapienza" - DAI Ematologia, Rome
  - Humanitas, Rozzano
  - Ospedale Maggiore San Giovanni Battista, Torino
  - Ospedale di Circolo Fondazione Macchi, Varese
- Clinic Hospital Universitari, Barcelona, Spain
- IOSI, Bellinzona, Switzerland
- United Kingdom (2):
  - Barts & the London NHS Trust, London
  - Royal Marsden NHS Foundation Trust, London

REFERENCES:
- [Derived] Ceriani L, Milan L, Martelli M, Ferreri AJM, Cascione L, Zinzani PL, Di Rocco A, Conconi A, Stathis A, Cavalli F, Bellei M, Cozens K, Porro E, Giovanella L, Johnson PW, Zucca E. Metabolic heterogeneity on baseline 18FDG-PET/CT scan is a predictor of outcome in primary mediastinal B-cell lymphoma. Blood. 2018 Jul 12;132(2):179-186. doi: 10.1182/blood-2018-01-826958. Epub 2018 May 2. PMID 29720487
- [Derived] Ceriani L, Martelli M, Zinzani PL, Ferreri AJ, Botto B, Stelitano C, Gotti M, Cabras MG, Rigacci L, Gargantini L, Merli F, Pinotti G, Mannina D, Luminari S, Stathis A, Russo E, Cavalli F, Giovanella L, Johnson PW, Zucca E. Utility of baseline 18FDG-PET/CT functional parameters in defining prognosis of primary mediastinal (thymic) large B-cell lymphoma. Blood. 2015 Aug 20;126(8):950-6. doi: 10.1182/blood-2014-12-616474. Epub 2015 Jun 18. PMID 26089397
- [Derived] Martelli M, Ceriani L, Zucca E, Zinzani PL, Ferreri AJ, Vitolo U, Stelitano C, Brusamolino E, Cabras MG, Rigacci L, Balzarotti M, Salvi F, Montoto S, Lopez-Guillermo A, Finolezzi E, Pileri SA, Davies A, Cavalli F, Giovanella L, Johnson PW. [18F]fluorodeoxyglucose positron emission tomography predicts survival after chemoimmunotherapy for primary mediastinal large B-cell lymphoma: results of the International Extranodal Lymphoma Study Group IELSG-26 Study. J Clin Oncol. 2014 Jun 10;32(17):1769-75. doi: 10.1200/JCO.2013.51.7524. Epub 2014 May 5. PMID 24799481